CLINICAL TRIAL: NCT00982202
Title: Pioglitazone in Alzheimer Disease Progression
Brief Title: Pioglitazone in Alzheimer Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: David Geldmaher, MD, University of Virginia Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0168; 1R01AG018905 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer Disease
Keywords: PPAR-gamma; inflammation
MeSH Terms: conditions — Alzheimer Disease; Inflammation | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PGZ (Experimental)
  Interventions: Drug: pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pioglitazone — 15mg tablet daily, increase by one pill at one-week intervals based on reported tolerability; maintain best tolerated dose (1 to 3 tablets daily) for ~18months
  Other Names: Actos
  Arms: PGZ
Drug: Placebo — 1 to 3 tablets daily for ~18 months
  Arms: Placebo

SUMMARY:
This study was designed to assess the safety and tolerability of pioglitazone, an approved drug for type 2 diabetes, in non diabetic patients with Alzheimer's disease. It was also designed to generate preliminary information on whether pioglitazone might slow progression of Alzheimer's disease.

DETAILED DESCRIPTION:
Inflammatory processes are important in the progressive loss of memory and thinking skills in Alzheimer's disease (AD). Laboratory studies show that drugs that bind to a protein known as "Peroxisome Proliferator Activated Receptor-gamma (PPARgamma)" act to reduce inflammatory responses in brain cells known as microglia when they are exposed to amyloid peptide, a major part of AD pathology. Therefore, drugs that activate PPARgamma have great potential for reducing the progression of AD. Pioglitazone (PGZ) activates PPARgamma and has shown favorable clinical experiences and safety profiles in patients with diabetes. This is a pilot study to determine the safety and tolerability of PGZ in patients with AD. Another goal of the study is to assess how clinical measures of cognition, daily function, and behavior might respond to PGZ treatment.

ELIGIBILITY:
Inclusion Criteria:

* CT or MRI since disease onset excluding structural lesions sufficient to account for the participant's dementia
* Mini-Mental State Exam (MMSE) score between 12 and 26, inclusively
* Clinical Dementia Rating (CDR) score of 1 or 2 (mild to moderate AD severity) at both screening and baseline
* Women must be 2-years post-menopausal or surgically sterile.
* Generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane); vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures
* Concomitant medications: Participants may be on stable doses of cholinesterase inhibitors for 90 days prior to screening (may not be started during the trial); antidepressant or antipsychotic medications are acceptable if symptoms are controlled and therapy is at stable dosage for at least 30 days prior to screening; vitamin E at 200 IU daily will be provided to all participants beginning at baseline/randomization (higher doses must be discontinued at the screening visit)

Exclusion Criteria:

* Absence of a reliable caregiver who is willing to participate and comply with protocol responsibilities
* Diabetes mellitus requiring medical therapy (diet-controlled diabetes is acceptable)
* Acute or chronic liver failure, hepatitis within the last two years, or history of drug-induced liver transaminase elevations
* Heart failure meeting New York Heart Association Grade III or IV criteria (i.e., functionally disabling)
* Evidence of active gastrointestinal, renal, pulmonary, endocrine or cardiovascular system disease sufficient to cause cognitive impairment or interfere with past levels of daily function; participants with controlled hypertension (supine diastolic BP < 95mmHg), right bundle branch block (complete or partial) and pacemakers may be included in the study; participants with thyroid disease also may be included in the study, provided they are euthyroid on treatment
* Active treatment for cancer or history of cancer within 3 years of screening (basal cell and squamous cells skin cancers are acceptable; incidental finding of carcinoma cells at transurethral prostate resection without subsequent medical or surgical therapy is acceptable)
* Evidence of other psychiatric/neurologic disorders sufficient to be the primary source of cognitive impairment (i.e., stroke, idiopathic Parkinson's disease, schizophrenia, bipolar or unipolar depression, seizure disorder, head injury with loss of consciousness within the past year) or a modified Hachinski's ischemia score of 5 or greater; delusions, hallucinations or depression not successfully treated or not on stable medical therapy for these conditions 30 days prior to enrollment; known or suspected history (within the past 10 years) of alcoholism or drug misuse
* Participants and/or caregivers who are unwilling or unable to fulfill the requirements of the study
* Any condition which would make the participant or the caregiver, in the opinion of the investigator, unsuitable for the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | baseline, monthly for 1 year, then 15 and 18 months

SECONDARY OUTCOMES:
Laboratory abnormalities | baseline, monthly for 1 year, then 15 and 18 months
Cognition | baseline, 3, 6, 9, 12, 15, and 18 months
Activities of Daily Living (ADL) | baseline, 3, 6, 9, 12, 15, and 18 months
Behavior | baseline, 3, 6, 9, 12, 15, and 18 months
Global function | baseline, 3, 6, 9, 12, 15, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Geldmaher, MD, Principal Investigator — University of Virginia Health System
Locations (2):
- United States (2):
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Heneka MT, Sastre M, Dumitrescu-Ozimek L, Hanke A, Dewachter I, Kuiperi C, O'Banion K, Klockgether T, Van Leuven F, Landreth GE. Acute treatment with the PPARgamma agonist pioglitazone and ibuprofen reduces glial inflammation and Abeta1-42 levels in APPV717I transgenic mice. Brain. 2005 Jun;128(Pt 6):1442-53. doi: 10.1093/brain/awh452. Epub 2005 Apr 7. PMID 15817521
- [Background] Jiang Q, Heneka M, Landreth GE. The role of peroxisome proliferator-activated receptor-gamma (PPARgamma) in Alzheimer's disease: therapeutic implications. CNS Drugs. 2008;22(1):1-14. doi: 10.2165/00023210-200822010-00001. PMID 18072811
- [Background] Lincoff AM, Wolski K, Nicholls SJ, Nissen SE. Pioglitazone and risk of cardiovascular events in patients with type 2 diabetes mellitus: a meta-analysis of randomized trials. JAMA. 2007 Sep 12;298(10):1180-8. doi: 10.1001/jama.298.10.1180. PMID 17848652
- [Derived] Geldmacher DS, Fritsch T, McClendon MJ, Landreth G. A randomized pilot clinical trial of the safety of pioglitazone in treatment of patients with Alzheimer disease. Arch Neurol. 2011 Jan;68(1):45-50. doi: 10.1001/archneurol.2010.229. Epub 2010 Sep 13. PMID 20837824